CLINICAL TRIAL: NCT04596488
Title: Pharmacodynamics of Efavirenz 400mg in Treatment-naïve Chinese HIV-infected Patients in a Prospective Cohort Study
Brief Title: Efavirenz 400mg in Treatment-naïve Chinese HIV-infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: National Key Technologies R&D Program for the 13th Five-year Plan (Unknown); National Key Technologies R&D Program for the 12th Five-year Plan (Unknown); CAMS Initiative for Innovative Medicine (Unknown)
Responsible Party: Principal Investigator, LI Taisheng, Director in department of Infectious Diseases, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XL001
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: HIV-1-infection
Keywords: Efavirenz 400mg; Chinese HIV-infected patients
MeSH Terms: interventions — efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Efavirenz 400mg+TDF+3TC (Experimental): Combined antiretroviral therapy(cART) consisting of three regimens such as efavirenz, tenofovir and lamivudine is an effective measure for the treatment of HIV-1 infection.Efavirenz 600mg daily was approved by the US Food and Drug Administration in 1998. In this single-arm research, patients were treated with a reduced 400mg dose of efavirenz combined with tenofovir 300mg and lamivudine 300mg once a day. This treatment had to be maintained indefinitely due to the existence of HIV reservoir.
  Interventions: Drug: Efavirenz 400mg

INTERVENTIONS:
Drug: Efavirenz 400mg — HIV-infected patients were treated with efavirenz 400mg combined with tenofovir 300mg and lamivudine 300mg.

SUMMARY:
Evaluating the efficacy, pharmacodynamics, and safety of Efavirenz 400mg in treatment-naïve Chinese HIV-infected patients.

DETAILED DESCRIPTION:
Treatment-naive HIV-infected patients are designed to enroll and receive efavirenz 400mg combined with tenofovir (TDF) and lamivudine (3TC) as initial antiretroviral regimens, and monitoring for 48 weeks, to evaluate efavirenz concentration, T-cell subsets, HIV RNA load, and neuropsychiatric tests with Hamilton depression scale (HAMD) and Pittsburgh sleep quality index (PSQI) at baseline, 4, 12, 24, 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* (1) HIV treatment-naïve, (2) age between 18 years or older, (3) be willing to complete the HAMD and PSQI scale and follow-up regularly, (5) not participating in other studies.

Exclusion Criteria:

* (1) acute HIV-1-infected patients, (2) an AIDS-defining illness such as pneumocystis pneumonia, tuberculosis within 2 weeks of entry, (3) transaminase and alkaline phosphatase levels beyond three times the upper limit of the normal range, bilirubin level more than 2.5 times the upper limit of the normal range, and serum creatinine level excess 1.5 times the upper limit of the normal range, (4) pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Viral suppression | 48 weeks
  The proportion of patients with viral load less than 50 copies/mL

SECONDARY OUTCOMES:
Drug concentration | 48 weeks
  The proportion of patients with plasma efavirenz concentration between 1 mg/L and 4mg/L
Neuropsychiatric adverse events | 48 weeks
  The proportion of patients with HAMD <8 and PSQI <10 (less neuropsychiatric adverse effects)

CONTACTS AND LOCATIONS:
Overall Officials: Taisheng Li, MD, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu L, Peng W, Song X, Li Y, Han Y, Zhu T, Fu Q, Du X, Cao W, Li T. Pharmacodynamics of efavirenz 400 mg in treatment-naive Chinese HIV-infected patients in a prospective cohort study. BMC Infect Dis. 2021 Jan 23;21(1):112. doi: 10.1186/s12879-021-05802-8. PMID 33485301